CLINICAL TRIAL: NCT00559780
Title: Muscle Function in the Elderly After Hip-Replacement Surgery - Effects of Long Term Disuse and Physical Training
Brief Title: Muscle Function in Elderly Postoperative Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKF:01058/00; HKF:01058/00
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Rehabilitation Strategies for Elderly Post-Operative Patients
Keywords: Resistance training; Aging; hip-surgery
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 12 weeks of resistance training
  Interventions: Behavioral: Resistance training
- 2 (Experimental): 12 weeks of neuromuscular electrical stimulation
  Interventions: Behavioral: Neuromuscular electrical stimulation of the quadriceps muscle
- 3 (Other): 12 weeks of standard rehabilitation
  Interventions: Behavioral: Standard rehabilitation

INTERVENTIONS:
Behavioral: Resistance training — 12 weeks of resistance training (3/week)
  Arms: 1
Behavioral: Neuromuscular electrical stimulation of the quadriceps muscle — 12 weeks of neuromuscular electrical stimulation of the quadriceps muscle (1h/day)
  Arms: 2
Behavioral: Standard rehabilitation — 12 weeks of standard physiotherapy exercises (1h/day)
  Arms: 3

SUMMARY:
During the last decades there has been an increase in the relative proportion and life expectancy of elderly people in the industrialised countries. Consequently the amount of elderly with diseases and disabilities related to aging has increased. It therefore appears paramount to gain a better understanding of how disuse and immobilisation affects neuromuscular properties in the elderly, as well as to identify training regimes that ensures an effective rehabilitation.The population of interest in the present study was elderly individuals with long term hip-osteoarthritis undergoing a hip-replacement operation. The study was divided in two parts, a cross-sectional study and an intervention study.

The cross-sectional study investigated muscle size, maximal muscle strength, specific force, neural drive and explosive muscle force characteristics in elderly individuals who were affected by unilateral prolonged disuse due to hip-osteoarthritis. The data clearly indicated that the side with hip-osteoarthritis was affected by a marked decrease in muscle mass, maximal muscle strength, neural drive and explosive muscle force characteristics compared to the unaffected side.

The intervention study investigated if elderly patients that undergo hip-replacement surgery could benefit from additional training in the early postoperative phase. The data clearly demonstrated that resistance training was an effective and safe way to increase muscle mass, maximal muscle strength, neuromuscular activity, functional performance and decrease the hospitalisation period compared to regimes of conventional rehabilitation regimen or electrical muscle stimulation. Additionally the intervention study demonstrated that resistance training effectively induced marked increases in explosive muscle force characteristics in elderly subjects compared to rehabilitation regimes using electrical muscle stimulation or conventional rehabilitation. Furthermore, the gains in maximal muscle strength and explosive muscle force characteristics were accompanied by significant increases in EMG amplitudes. Furthermore, the demonstration that explosive muscle force capacity of the neuromuscular system remains trainable in elderly recovering from prolonged limb disuse and major surgery may have important implications for future rehabilitation programs, especially when considering the importance of rapid muscle force capacity on postural balance, maximal walking speed and other tasks of daily life actions.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years
* Unilateral primary hip replacement due to hip osteoarthritis in patients

Exclusion Criteria:

* Cardiopulmonary, neurological or cognitive problems

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-05; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suetta, MD, PhD, Principal Investigator — Institute of Sports Medicine copenhagen, Bispebjerg Hospital
Locations (1):
- Institute of Sports Medicine, Bispebjerg Hospital, Copenhagen, Denmark